CLINICAL TRIAL: NCT00403520
Title: Assessment of the Comparative Effect of Donepezil 10mg/d and Placebo on Clinical and Radiological Markers in Patients With Mild Cognitive Disorders
Brief Title: Hippocampus Study: Comparative Effect of Donepezil 10mg/d and Placebo on Clinical and Radiological Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-E033-415
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Mild cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Experimental 1 (Experimental)
  Interventions: Drug: Experimental 1
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Experimental 1 — Drug: Donepezil Hydrochloride 10 mg orally for 12 months
  Arms: Experimental 1
Drug: Placebo Comparator — Drug: Placebo Matching placebo orally for 12 months
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to demonstrate that donepezil slows the progression of Alzheimer's disease (AD) using magnetic resonance imaging (MRI) of the brain to measure the volume of the hippocampus in patients with pre-dementia Alzheimer's disease.

DETAILED DESCRIPTION:
The development of a new automated method of measurement of the volume of the hippocampus allows confirming these results in patients presenting with pre-dementia Alzheimer's Disease (AD), treated with donepezil in order to verify if this product is capable of stopping the speed of the atrophy of the hippocampus in patients and more specifically in those who will evolve to AD, compared to a placebo. This method is a semi automatic segmentation of the hippocampus from MRI, made by competitive region growing.

It was developed at the cognitive neurosciences and MRI laboratory in Pitié-Salpêtrière hospital. This method was validated on healthy subjects and Alzheimer's disease patients by comparison with manual segmentation.

Neuropsychological tests will be realized in order to supervise the clinical evolution of the patients and to correlate these results to the progression of the atrophy of the hippocampus.

ELIGIBILITY:
Inclusion Criteria (Baseline Visit ("V0"):

1.Men or Women 50 years old or more. 2. Patients with mild cognitive impairment (MCI) with progressive hippocampal amnestic syndrome, isolated or associated to other cognitive disorders defined by the Free and cued selective reminding test ( FCSRT ) with Free Recall < or = 17 OR Total Recall < 40 , according to the Grober and Buschke procedure, modified according to the results of PREAL study 3.Clinical Dementia Rating (CDR) = 0.5 4. General cognition and functional performance sufficiently preserved such that a diagnosis of Possible or Probable Alzheimer's Disease based on Diagnostic and Statistical Manual of Mental Disorders DSM-IV criteria) cannot be made by the site physician at the time of the screening visit. This evidence must be fully documented in the subject's study file before the Randomization visit.

5. Outpatient with an informant person: person from his/her close circle having a regular weekly contact with the patient and accepting to answer to assessment questionnaires.

6. Visual, hearing capacities (authorized equipment) and oral or written expression, sufficient for the correct performance of the tests (according to the physician's opinion).

7. Patient and informant person having signed the written informed consent form.

Exclusion Criteria (Baseline Visit ("V0"):

1. Patients with a contraindication to MRI:

   * Pacemaker, cardiac defibrillator or neurostimulator wearers
   * Wearers of implanted material activated by an electric, magnetic or mechanical system
   * Wearers of haemostatic clips of intracerebral aneurysms or carotid arteries
   * Wearers of cochlear implants
   * Patients with an intraocular metallic foreign body
   * Claustrophobic patients
   * Any other contra-indication to MRI
2. Patients with an evolutive psychiatric pathology and/or unstable according to DSM-IV, particularly:

   * Major depressive episode during the previous 2 years or recurrent depression or bipolar disorders according to the DSM-IV and/or score >= 12 according to the 17-items depressive Hamilton's Scale
   * Patients presenting early hallucinations or cognitive fluctuations
3. Patients with neurological disorders:

   * Partial complex epilepsy
   * Dementia of any origin
   * Patients with Parkinson's disease
4. Any patient with a history of an intercurrent lesion found in brain imaging studies.
5. Patient presenting a major repercussion on the autonomy, assessed by Instrumental Activities of Daily Living (IADL) Lawton score higher or equal to 2 in at least 2 items or higher than 2 in at least 1 item, confirmed by an informant person.
6. Patient having less than 14 words at the identification phase of the FCSRT (Free and Cued Selective Reminding Test)
7. Known vitamin B12 or folates deficiency (except if replacement treatment of stable posology since at least 6 months before selection) or known syphilis.
8. Abnormal Thyroid function (T3, T4, ultrasensitive thyroid stimulating hormone (TSH). Euthyroid patients treated with stable doses for at least 3 months could be included.
9. Insulin dependent diabetes or diabetes not controlled by a regimen and/or oral antidiabetics, obstructive pulmonary disease, unstable asthma, recent hematological and/or oncological disorders (2 years).
10. Gastrointestinal, renal, hepatic, endocrine or cardiovascular clinically significant disease. Atrioventricular block of 2nd or 3rd degree on ECG.
11. Patient with bradycardia < or = 50 beats per minute.
12. Patient with unstable hypertension (systolic blood pressure > 160 mmHg and /or diastolic blood pressure > 95 mmHg) assessed by the investigator, the patient being treated or not by antihypertensive drugs.
13. Patient previously treated with central cholinesterase inhibitors or memantine whatever the duration of the treatment and the date of prescription
14. Patient treated by a non-authorized drug during the study
15. Known or suspected history (5 years) of alcoholism, or abusive drug use.
16. Patients with known hypersensitivity to donepezil chlorhydrate, to piperidine derivatives or to one of the excipients of the drug.
17. Patients having participated in a clinical trial during the previous 3 months.

Inclusion criteria (Visit 1):

1. Patients with mild cognitive impairment (MCI) with progressive hippocampal amnestic syndrome, isolated or associated to other cognitive disorders
2. General cognition and functional performance sufficiently preserved such that a diagnosis of Possible or Probable Alzheimer's Disease based on clinical and neuro-imaging findings (NINCDS-ADRDA or DSM-IV criteria) cannot be made by the site physician at the time of the screening visit. This evidence must be fully documented in the subject's study file.
3. Outpatient with an informant person: person from his/her close circle having a regular weekly contact with the patient and accepting to answer to assessment questionnaires
4. Patients having performed an electrocardiogram (ECG) within the previous 6 months
5. Visual, hearing capacities (authorized equipment) and oral or written expression, sufficient for the correct performance of the tests (according to the physician's opinion)
6. Clinical laboratory values must be within normal limits, or if abnormal, judged clinically insignificant by the investigator (not likely to cause cognitive impairment or medical instability)
7. Clinical Dementia Rating (CDR - sum of the boxes) = 0.5

Exclusion criteria (Visit 1):

1. Patients with an evolutive psychiatric pathology and/or unstable according to DSM-IV, particularly:

   * Major depressive episode ongoing or recurrent depression or bipolar disorders according to the DSM-IV and/or score >or = 12 according to the 17-items depressive Hamilton's Scale
   * Patients presenting early hallucinations or cognitive fluctuations
2. Any patient presenting with an intercurrent lesion in MRI performed at screening must be excluded from the study, apart from minor non-progressive lesions not altering brain morphology
3. Patients with neurological disorders :

   * Partial complex epilepsy
   * Dementia of any origin
   * Patients with Parkinson's disease
4. Patient with One or more MRI Exclusion criteria :

   * Stroke sequelae
   * More than one ischemic lacuna
   * Age related white matter changes on Flair images >Fazekas and Schmidt grade 2
   * Active ischemic lesion on Diffusion weighted Images (DWI)
5. Patient presenting a major repercussion on the autonomy, assessed by IADL Lawton score higher or equal to 2 in at least 2 items or higher than 2 in at least 1 item, confirmed by an informant person.
6. Known vitamin B12 or folates deficiency (except if replacement treatment of stable posology since at least 6 months before selection) or known syphilis.
7. Abnormal Thyroid function (T3, T4, free thyroxine index, TSH). Euthyroid patients treated with stable doses for at least 3 months could be included.
8. Insulin dependent diabetes or diabetes not controlled by a regimen and/or oral antidiabetics, obstructive pulmonary disease, unstable asthma, recent hematological and/or oncological disorders (<= 2 years).
9. Gastrointestinal, renal, hepatic, endocrine or cardiovascular clinically significant disease. Atrioventricular block of 2nd or 3rd degree on ECG.
10. Patients with bradycardia <= 50.
11. Patients with unstable hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 95mmHg) assessed by the investigator, the patient being treated or not by anti hypertensive drugs.
12. Patient previously treated with central cholinesterase inhibitors or memantine whatever the duration of the treatment and the date of prescription
13. Patient treated by a non-authorized drug during the study
14. Known or suspected history (<= 5 years) of alcoholism, or abusive drug use.
15. Patients with known hypersensitivity to donepezil chlorhydrate, to piperidine derivatives or to one of the excipients of the drug.
16. Patients having participated in a clinical trial during the previous 3 months.
17. Patient treated by a non-authorized drug during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-11; Primary Completion 2008-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Evolution of the volume of the Hippocampi, measured by magnetic resonance imaging (MRI), between D0 and final visit (12 months ). | ( Day 0 to 12 months or in case of premature withdrawal after 6 months period

SECONDARY OUTCOMES:
Evolution of the neuropsychological scores between Day 0 and final visit. | Day 0 to 12 during treatment and at 18 months follow up
  Outcome Measure Description: Patients will perform neuropsychological and independence tests including (16 items free recall/cued recall test using the Grober-Buschke method, Mini-Mental State Examination (MMSE), Clinical Dementia Rating (CDR) sum of the boxes and Instrumental Activities of Daily Living (IADL), and will be evaluated using the Hamilton Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Tonelli, Study Director — Eisai France
Locations (1):
- CHU Gui de Chauliac, Montpellier, France

REFERENCES:
- [Derived] Diaz-Galvan P, Lorenzon G, Mohanty R, Martensson G, Cavedo E, Lista S, Vergallo A, Kantarci K, Hampel H, Dubois B, Grothe MJ, Ferreira D, Westman E. Differential response to donepezil in MRI subtypes of mild cognitive impairment. Alzheimers Res Ther. 2023 Jun 23;15(1):117. doi: 10.1186/s13195-023-01253-2. PMID 37353809
- [Derived] Cavedo E, Dubois B, Colliot O, Lista S, Croisile B, Tisserand GL, Touchon J, Bonafe A, Ousset PJ, Rouaud O, Ricolfi F, Vighetto A, Pasquier F, Galluzzi S, Delmaire C, Ceccaldi M, Girard N, Lehericy S, Duveau F, Chupin M, Sarazin M, Dormont D, Hampel H; Hippocampus Study Group. Reduced Regional Cortical Thickness Rate of Change in Donepezil-Treated Subjects With Suspected Prodromal Alzheimer's Disease. J Clin Psychiatry. 2016 Dec;77(12):e1631-e1638. doi: 10.4088/JCP.15m10413. PMID 27780331
- [Derived] Teipel SJ, Cavedo E, Grothe MJ, Lista S, Galluzzi S, Colliot O, Chupin M, Bakardjian H, Dormont D, Dubois B, Hampel H; Hippocampus Study Group. Predictors of cognitive decline and treatment response in a clinical trial on suspected prodromal Alzheimer's disease. Neuropharmacology. 2016 Sep;108:128-35. doi: 10.1016/j.neuropharm.2016.02.005. Epub 2016 Feb 10. PMID 26876309